CLINICAL TRIAL: NCT01121874
Title: Suture Fixation System Versus Tendonous Reconstruction in Thumb Carpometacarpal Arthroplasty: a Randomized Controlled Trial
Brief Title: Suture Fixation System Versus Tendonous Reconstruction in Carpometacarpal (CMC) Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J&M Shuler (Industry)
Responsible Party: Principal Investigator, Michael Shuler, Hand and Upper Extremity Specialist, J&M Shuler
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMC-101
Record Dates: First submitted 2010-04-09; First posted 2010-05-12 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Thumb Carpometacarpal Arthritis
Keywords: CMC arthritis; thumb carpometacarpal arthritis; basal joint arthritis; thumb CMC arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LRTI (Active Comparator): These patients will undergo ligament reconstruction with tendon interposition (LRTI) surgery. They will serve as a control group, against which to compare the investigational surgical technique.
  Interventions: Procedure: Ligament Reconstruction with Tendon Interposition (LRTI)
- Suture fixation system (Experimental): CMC arthroplasty which reconstructs palmar oblique ligament using a suture fixation system.
  Interventions: Procedure: Ligament reconstruction with suture fixation system
- Suture fixation system + 2 week immobilization (Experimental): CMC arthroplasty which reconstructs palmar oblique ligament using a suture fixation system, and with a decreased immobilization time from 6 to 2 weeks post-surgery.
  Interventions: Procedure: Ligament reconstruction with suture fixation system

INTERVENTIONS:
Procedure: Ligament reconstruction with suture fixation system — CMC arthroplasty consisting of reconstruction of the palmar oblique ligament using a suture fixation system
  Other Names: Arthrex Mini TightRope
  Arms: Suture fixation system
Procedure: Ligament Reconstruction with Tendon Interposition (LRTI) — commonly performed CMC arthroplasty technique, consisting of a trapeziectomy, followed by palmar oblique ligament reconstruction using a harvested flexor tendon from the wrist.
  Arms: LRTI
Procedure: Ligament reconstruction with suture fixation system — CMC arthroplasty consisting of reconstruction of the palmar oblique ligament using a suture fixation system, with a decreased period of immobilization from 6 weeks to 2 weeks.
  Other Names: Arthrex Mini TightRope
  Arms: Suture fixation system + 2 week immobilization

SUMMARY:
Thumb carpometacarpal (CMC) arthritis affect 1 in 4 females and 1 in 12 males. Patients who fail to respond to conservative treatment may benefit from surgery; however, controversy exists over the most effective surgical technique. A popular technique, ligament reconstruction with tendon interposition (LRTI) involves a trapeziectomy, followed by reconstruction of the palmar oblique ligament using a harvested flexor tendon from the wrist.

We believe that use of a suture fixation system to reconstruct the palmar oblique ligament, instead of harvesting a wrist tendon, may provide a superior repair. The objective of this study is to compare functional outcome measurements among patients who receive CMC arthroplasty using a suture fixation system (investigational group) to those who receive LRTI surgery (control group). We hypothesize that patients in the investigational group will demonstrate superior functionality, compared to patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >18.
* Eaton Stage III or IV CMC arthritis
* Failure to respond to conservative treatment

Exclusion Criteria:

* Previous surgical interventions on that thumb
* Upper extremity neurological dysfunction
* Inability to effectively communicate with the research staff, due to hearing impairment, cognitive impairment, or a language barrier
* Unwilling or unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04-12 (Actual); Primary Completion 2012-05-21 (Actual); Study Completion 2012-07-25 (Actual)

PRIMARY OUTCOMES:
Overall functionality | Baseline
  Functionality will be assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, which assesses functionality of the upper extremity, and Short Form 36 (SF-36) health outcomes assessment, which quantifies global functionality (not specific to the upper extremity).
Overall Functionality | 6 wks
Overall Functionality | 3 mos
Overall Functionality | 6 mos
Overall Functionality | 12 months
Overall Functionality | 24 months

SECONDARY OUTCOMES:
Analog pain scale | Baseline, 2 wks, 6 wks, 3 mos, 6 mos, 12 mos, 24 mos
  Pain will be assessed using the visual analog pain scale, which asks the patient to rate their pain on a scale from 1 to 10.
Strength measures | Baseline, 6 wks, 3 mos, 6 mos, 12 mos, 24 mos
  Strength will be assessed via key and tip pinch strength and grip strength, using a dynamometer
Range of motion | Baseline, 6 wks, 3 mos, 6 mos, 12 mos, 24 mos
  Range of motion (ROM) will be assessed via radial and palmar abduction (degrees) and opposition (cm).
Operative time | Baseline, 6 wks, 3 mos, 6 mos, 12 mos, 24 mos
  Operative time in minutes
Scaphometacarpal distance | Baseline, 6 wks, 3 mos, 6 mos, 12 mos, 24 mos
  Distance between the distal pole of the scaphoid and the proximal aticular surface of the metacarpal. Taken in stressed and relaxed views

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shuler, MD, Principal Investigator — Athens Orthopedic Clinic, PA
Locations (1):
- Athens Orthopedic Clinic, Athens, Georgia, United States